CLINICAL TRIAL: NCT03769558
Title: Supplemental Data for the Juvenile Idiopathic Arthritis FDA Written Request
Brief Title: A Study of Juvenile Idiopathic Arthritis Patients Given Abatacept and the Number of Infections or Malignancies That Occur
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM101-643
Record Dates: First submitted 2018-12-06; First posted 2018-12-07 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- JIA patients prescribed abatacept
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — Non-Interventional

SUMMARY:
This study will determine the incidences of infections and malignancies among JIA patients treated with abatacept

ELIGIBILITY:
Inclusion Criteria:

* Two diagnoses of JIA (ICD-9 code 714.3x) within 90 days
* Age less than 18 years at the time of second of the two diagnoses
* Index date is the date of initiating treatment with abatacept

Exclusion Criteria:

* Greater than or equal to 18 years of age

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include all patients with JIA who are treated with abatacept
Sampling Method: Probability Sample
Enrollment: 264 (Actual)
Dates: Start 2016-07-12 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Incidence of infections | 110 months

SECONDARY OUTCOMES:
Incidence of malignancies | 110 months

CONTACTS AND LOCATIONS:
Locations (1):
- Local Institution, Princeton, New Jersey, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm